CLINICAL TRIAL: NCT03518268
Title: The Efficacy of the Probiotic Supplement Vivomixx on Prevention of Bone Loss in Early Menopausal Women With Breast Cancer Treated With an Aromatase Inhibitor
Brief Title: Vivomixx for Prevention of Bone Loss in Women With Breast Cancer Treated With an Aromatase Inhibitor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Perrigo Company (Industry)
Responsible Party: Principal Investigator, michal roll, Deputy Director General for R&D, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0124-18-TLV
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Osteoporosis, Osteopenia
Keywords: probiotics; aromatase inhibitors; bone mass; postmenopausal
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dietary supplement Vivomixx (Active Comparator): Vivomixx sachets contains a mixture of 450 billion viable lyophilized bacteria from 8 strains: Lactobacillus paracasei DSM 24733, Lactobacillus plantarum DSM 24730, Lactobacillus acidophilus DSM 24735, Lactobacillus delbrueckii subspecies bulgaricus DSM 24734, Bifidobacterium longum DSM 3 24736, Bifidobacterium infantis DSM 24737, Bifidobacterium breve DSM 24732, and Streptococcus thermophilus DSM 24731
  Interventions: Drug: Vivomixx
- Placebo (Placebo Comparator): The placebo sachets contain the inactive ingredients maltose and silicon dioxides
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vivomixx — The intervention consists of 2 sachets a day containing the probiotic Vivomixx, for 6 months
  Arms: Dietary supplement Vivomixx
Drug: Placebo — The intervention consists of 2 sachets a day of placebo, for 6 months
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of the probiotic food supplement Vivomixx in the prevention of bone loss occurring in post menopausal women with breast cancer treated with an aromatase inhibitor. Half of the participants will receive Vivomixx while the other half will receive a placebo. The primary endpoint is to assess changes of bone turnover markers during the period of 6 months.

DETAILED DESCRIPTION:
Aromatase inhibitors function to reduce estrogen levels. They are considered first-line treatment for postmenopausal women with estrogen receptor-positive breast cancer. Estrogen depletion leads to significant loss of bone mineral density and an increased fracture risk. One contributing mechanism to "estrogen deficiency associated bone loss" is the increase in systemic and local gut inflammatory responses upon estrogen deficiency. Probiotics have been shown to decrease inflammatory cytokine formation in both the systemic circulation and gut.

Vivomixx is a high potency probiotic medical food designated for the dietary management of inflammatory gut conditions in adults and children and is currently being studied in clinical trials in a wide variety of inflammatory conditions such as asthma and diabetes. In preclinical studies Vivomixx has been shown to protect from estrogen deficient bone loss.

ELIGIBILITY:
Inclusion criteria

1. Age≥ 35 years
2. Breast cancer stages 1-3 (non metastatic)
3. Under treatment with aromatase inhibitors
4. In menopausal status for ≤10y
5. Estrogen receptor positive tumor
6. CTX ≥300 pg/ml

Exclusion criteria

1. Distant metastases
2. Additional active primary malignancy
3. Metabolic bone disease (primary hyperparathyroidism, hyperthyroidism, paget, osteomalacia etc)
4. Glucocorticoid treatment (chronic or high dose >7.5 mg in the last three months)
5. Bisphosphonate treatment for more than 3 months in the last 2 years
6. Bone densitometry (DXA) T-Score <-2 unless not a candidate for antiresorptive therapy (unwilling/unable to take treatment)
7. Lactose intolerant subjects

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Collagen type 1 cross-linked C-telopeptide (CTX) | 3-6 months
  Change in percent in CTX in serum compared to placebo
Serum type 1 procollagen (N-terminal) P1NP | 3-6 months
  Change in percent in serum in P1NP compared to placebo

SECONDARY OUTCOMES:
Alkaline phosphatase/ bone specific alkaline phosphatase | 3-6 months
  Change in percent in alkaline phosphatase/ bone specific alkaline phosphatase in serum compared to placebo
Osteocalcin | 3-6 months
  Change in percent in osteocalcin in serum compared to placebo
Sclerostin | 3-6 months
  Change in percent in sclerostin in serum compared to placebo
Tumor-necrosis factor-alpha | 3-6 months
  Change in percent in tumor-necrosis factor-alpha in serum compared to placebo
Interleukin-17 | 3-6 months
  Change in percent in interleukin-17 in serum compared to placebo
Receptor activator of nuclear factor kappa B ligand (RANK-ligand) | 3-6 months
  Change in percent in RANK-ligand in serum compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Naftali Stern, M.D, Study Director — Tel-Aviv Sourasky Medical Center